CLINICAL TRIAL: NCT04625101
Title: Phase 2 Multicenter, Randomized, Double-Blind, Placebo-Controlled, Parallel-Group Study to Assess the Efficacy, Safety, Tolerability, and Pharmacokinetics of NBI-827104 in Pediatric Subjects With Epileptic Encephalopathy With Continuous Spike-and-Wave During Sleep
Brief Title: Efficacy, Safety, Tolerability, and Pharmacokinetics of NBI-827104 in Pediatric Subjects With Epileptic Encephalopathy With Continuous Spike-and-Wave During Sleep
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Neurocrine Biosciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NBI-827104-CSWS2010; 2020-003141-11 (EudraCT Number)
Record Dates: First submitted 2020-11-06; First posted 2020-11-12 (Actual); Results first posted 2025-09-05 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-09

CONDITIONS: Epileptic Encephalopathy; Continuous Spike and Wave During Sleep

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- NBI-827104 (Experimental): NBI-827104 administered orally for 13 weeks.
  Interventions: Drug: NBI-827104
- Placebo (Placebo Comparator): Placebo administered orally for 13 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: NBI-827104 — Triple T-type calcium channel blocker.
  Arms: NBI-827104
Drug: Placebo — Non-active dosage form.
  Arms: Placebo

SUMMARY:
This is a phase 2, double-blind study to assess the efficacy, safety, tolerability, and pharmacokinetics of NBI-827104 when administered once daily for 13 weeks in pediatric subjects with Epileptic Encephalopathy with Continuous Spike-and-Wave During Sleep (EECSWS).

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent by the parent(s) or legal representative(s) and, if applicable, assent from developmentally capable pediatric subjects.
2. Diagnosis of EECSWS.
3. Have diagnosis of EECSWS confirmed by the Diagnosis Confirmation Panel (DCP).
4. Stable dosage and stable time of intake of at least 1 and up to 3 antiseizure medications (ASMs) excluding systemic corticosteroids and intravenous immunoglobulin (IVIG), from 4 weeks prior to screening and anticipated to be stable from screening until end of study (EOS). Vagal nerve stimulator (VNS) and ketogenic diet are not counted as ASMs.
5. Treatment other than ASMs (excluding systemic corticosteroids and IVIG) must be at a stable dosage from 2 weeks prior to screening and anticipated to be stable from screening until EOS.

Exclusion Criteria:

1. Lennox-Gastaut syndrome, Doose syndrome (epilepsy with myoclonic-atonic seizures), or Dravet syndrome.
2. Presence of a relevant psychiatric disease interfering with cognitive or behavioral functioning (eg, depression, schizophrenia, autism spectrum disorder) unless associated with the EECSWS diagnosis as assessed by the investigator.
3. Presence of relevant neurological disorders other than EECSWS and its underlying conditions as judged by the investigator. Symptomatic conditions underlying EECSWS (eg, neonatal strokes) have to be stable for at least 1 year prior to screening.
4. Body weight <10 kg at randomization.
5. Clinically relevant findings in systolic blood pressure (SBP), diastolic blood pressure (DBP), or pulse rate at screening or Day 1 as determined by the investigator.
6. Have an average triplicate ECG corrected QT interval using Fridericia's formula (QTcF) >450 msec or presence of any significant cardiac abnormality at screening.
7. Clinically relevant findings in clinical laboratory tests (hematology, clinical chemistry including thyroid function parameters, and urinalysis) at screening as determined by the investigator.
8. Have aspartate aminotransferase (AST), alanine aminotransferase (ALT), or gamma-glutamyl transferase (GGT) levels >2 × the upper limit of normal (ULN) at screening.
9. Have mild to severe renal impairment as determined by the investigator.
10. Have taken cannabinoids, excluding Epidiolex®/Epidyolex®, within 30 days of screening.
11. Pulse therapy such as systemic corticosteroids and IVIG are prohibited for at least 8 weeks prior to screening.
12. Planned surgical intervention related to structural abnormalities of the brain from screening through the duration of the study.
13. Have received any other investigational drug within 30 days or 5 half-lives (if known), whichever is longer, of Day 1 or plan to use an investigational drug (other than the study treatment) during the study.
14. Any circumstances or conditions, which, in the opinion of the investigator, may affect full participation in the study or compliance with the protocol.

Ages: 4 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 24 (Actual)
Dates: Start 2021-04-26 (Actual); Primary Completion 2022-08-08 (Actual); Study Completion 2022-10-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Development Lead, Study Director — Neurocrine Biosciences
Locations (15):
- United States (8):
  - Neurocrine Clinical Site, Orange, California
  - Neurocrine Clinical Site, Aurora, Colorado
  - Neurocrine Clinical Site, Washington D.C., District of Columbia
  - Neurocrine Clinical Site, Miami, Florida
  - Neurocrine Clinical Site, Rochester, Minnesota
  - Neurocrine Clinical Site, Durham, North Carolina
  - Neurocrine Clinical Site, Cleveland, Ohio
  - Neurocrine Clinical Site, Philadelphia, Pennsylvania
- Neurocrine Clinical Site, Calgary, Alberta, Canada
- Neurocrine Clinical Site, Dianalund, Denmark
- Spain (2):
  - Neurocrine Clinical Site, Barcelona
  - Neurocrine Clinical Site, Madrid
- Switzerland (2):
  - Neurocrine Clinical Site, Basel
  - Neurocrine Clinical Site, Zurich
- Neurocrine Clinical Site, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- NBI-827104: NBI-827104 administered orally daily for up to 13 weeks.
- Placebo: Placebo administered orally daily for up to 13 weeks.
Period: Overall Study
Arm/Group | NBI-827104 | Placebo
Started | 16 | 8
Received at Least 1 Dose of Study Drug | 16 | 8
Full Analysis Set | 15 | 7
Completed | 15 | 7
Not Completed | 1 | 1
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Protocol Deviation | 1 | 0

BASELINE CHARACTERISTICS:
Population: Safety Analysis set included all participants who received at least one dose of study treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | NBI-827104 | Placebo | Total
Number analyzed (Participants) | 16 | 8 | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 16 | 8 | 24
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 3 | 10
  Male | 9 | 5 | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 0 | 3
  Not Hispanic or Latino | 13 | 8 | 21
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 15 | 7 | 22
  Race: Black or African American | 0 | 1 | 1
  Race: Other | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Ratio of Spike-Wave Index (SWI) During First Hour of Nonrapid Eye Movement (NREM) Sleep at Week 6
Description: The ratio of SWI at the end of Week 6 to baseline during the first hour (60 minutes) of NREM sleep based on centralized video-electroencephalograph (EEG) reading using a log base 10 scale. Baseline was defined as the last value measured prior to intake of study treatment on Day 1. SWI was defined as the percentage of seconds with ≥1 spike-wave complex(es) during defined periods of overnight NREM sleep.
Time Frame: Baseline to Week 6
Population: Full Analysis Set included all randomized participants who had at least 1 dose of study treatment and at least 1 efficacy video EEG assessment. The number of participants analyzed = the number of participants who were evaluable for this outcome measure.
Measure: Least Squares Mean (Standard Error); unit: Log-transformed ratio
Arm/Group | NBI-827104 | Placebo
Number analyzed (Participants) | 14 | 6
Log-transformed ratio | -0.02 (0.02) | 0.01 (0.04)
Statistical Analysis 1: Comparison: NBI-827104 vs Placebo; Test type: Superiority; p = 0.4326, ANCOVA

2. Secondary Outcome: Ratio of SWI During First Hour of NREM Sleep at Week 12
Description: The ratio of SWI at the end of Week 12 to baseline during the first hour (60 minutes) of NREM sleep based on centralized video-EEG reading using a log base 10 scale. Baseline was defined as the last value measured prior to intake of study treatment on Day 1. SWI was defined as the percentage of seconds with ≥1 spike-wave complex(es) during defined periods of overnight NREM sleep.
Time Frame: Baseline to Week 12
Population: Full Analysis Set included all randomized participants who had at least 1 dose of study treatment and at least 1 efficacy video EEG assessment.
Measure: Least Squares Mean (Standard Error); unit: Log-transformed ratio
Arm/Group | NBI-827104 | Placebo
Number analyzed (Participants) | 15 | 7
Log-transformed ratio | -0.05 (0.02) | 0.03 (0.03)

3. Secondary Outcome: Number of Participants Considered as Responders as Assessed by the Caregiver Global Impression of Change (CaGI-C) Score
Description: The CaGI-C is a 7-point scale that rates the caregiver's assessment of the overall improvement in the participants symptoms since the initiation of study treatment, ranging from 1 (very much improved) to 7 (very much worse). A responder was defined as a participant with a score of 1 (very much improved) or 2 (much improved).
Time Frame: Week 6 and Week 12
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | NBI-827104 | Placebo
Number analyzed (Participants) | 15 | 7
Participants
  Week 6 | 1 | 1
  Week 12 | 2 | 1

4. Secondary Outcome: Number of Participants Considered as Responders as Assessed by the Clinician Global Impression of Change (CGI-C) Score
Description: The CGI-C is a 7-point scale that rates the clinician's assessment of overall improvement in the participant's symptoms since the initiation of study treatment, ranging from 1 (very much improved) to 7 (very much worse). A responder was defined as a participant with a score of 1 (very much improved) or 2 (much improved).
Time Frame: Week 6 and Week 12
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | NBI-827104 | Placebo
Number analyzed (Participants) | 15 | 7
Participants
  Week 6 | 1 | 1
  Week 12 | 1 | 1

5. Secondary Outcome: Number of Participants Considered as Responders as Assessed by the Clinical Global Impression of Severity (CGI-S) Scores
Description: The CGI-S is a 7-point scale that rates the clinician's assessment of overall symptom severity, ranging from 1 (normal, not at all ill) to 7 (among the most extremely ill patients). A responder was defined as a participant with at least 1-point improvement in the CGI-S score from baseline.
Time Frame: Weeks 6 and 12
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | NBI-827104 | Placebo
Number analyzed (Participants) | 15 | 7
Participants
  Week 6 | 3 | 1
  Week 12 | 4 | 4

ADVERSE EVENTS:
Time Frame: Day 1 (after dosing) up to Week 17
Description: Safety analysis set included all randomized participants who had at least 1 dose of study treatment.
Arm/Group | NBI-827104 | Placebo
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/8
Serious Adverse Events (participants affected / at risk) | 1/16 | 0/8
Other Adverse Events (participants affected / at risk) | 11/16 | 8/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | NBI-827104 (N=16) | Placebo (N=8)
Seizure (Nervous system disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | NBI-827104 (N=16) | Placebo (N=8)
Flushing (Vascular disorders) | 1 | 0
Fatigue (General disorders) | 3 | 0
Pyrexia (General disorders) | 1 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Affect lability (Psychiatric disorders) | 2 | 0
Aggression (Psychiatric disorders) | 0 | 1
Depressed mood (Psychiatric disorders) | 1 | 0
Irritability (Psychiatric disorders) | 1 | 0
Restlessness (Psychiatric disorders) | 0 | 1
Suicidal ideation (Psychiatric disorders) | 0 | 1
Terminal insomnia (Psychiatric disorders) | 0 | 1
Alanine aminotransferase increased (Investigations) | 1 | 0
Blood creatine phosphokinase increased (Investigations) | 1 | 1
Blood triglycerides increased (Investigations) | 0 | 1
Lymphocyte count decreased (Investigations) | 1 | 0
Neutrophil count decreased (Investigations) | 2 | 0
Protein urine present (Investigations) | 0 | 1
White blood cell count decreased (Investigations) | 1 | 1
Vitamin D decreased (Investigations) | 0 | 1
Face injury (Injury, poisoning and procedural complications) | 0 | 1
Tachycardia (Cardiac disorders) | 1 | 0
Dizziness (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 2 | 0
Partial seizures (Nervous system disorders) | 1 | 0
Somnolence (Nervous system disorders) | 1 | 0
Tremor (Cardiac disorders) | 1 | 1
Eye pain (Eye disorders) | 0 | 1
Abdominal pain lower (Gastrointestinal disorders) | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 1 | 1
Haematochezia (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 1
Keratosis pilaris (Skin and subcutaneous tissue disorders) | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 1
Precocious puberty (Endocrine disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0
COVID-19 (Infections and infestations) | 2 | 2
Infection (Infections and infestations) | 1 | 0
Nasopharyngitis (Infections and infestations) | 0 | 1
Otitis media (Infections and infestations) | 1 | 0
Rash pustular (Infections and infestations) | 0 | 1
Suspected COVID-19 (Infections and infestations) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 1
Urinary tract infection (Infections and infestations) | 1 | 0
Viral infection (Infections and infestations) | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 3 | 1
Tremor (Nervous system disorders) | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2021-08-05): https://cdn.clinicaltrials.gov/large-docs/01/NCT04625101/Prot_000.pdf
  • Statistical Analysis Plan (2022-11-18): https://cdn.clinicaltrials.gov/large-docs/01/NCT04625101/SAP_001.pdf